CLINICAL TRIAL: NCT04237610
Title: Reward and Punishment Sensitivity in Bipolar Disorders
Acronym: Recodec-BP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC18.171; 2018-A01962-53 (Other: ID RCB)
Record Dates: First submitted 2020-01-10; First posted 2020-01-23 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Bipolar Disorder
Keywords: reinforcement learning
MeSH Terms: conditions — Bipolar Disorder | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bipolar disorder type I
  Interventions: Behavioral: behavioral assessment
- Bipolar disorder type II
  Interventions: Behavioral: behavioral assessment
- healthy controls
  Interventions: Behavioral: behavioral assessment

INTERVENTIONS:
Behavioral: behavioral assessment — Probabilistic learning task

SUMMARY:
Bipolar disorder (BD) represents a chronic mood disorder and one of the leading causes of disability worldwide. Complexity of its clinical presentations leads to delayed diagnosis and difficult management in routine clinical settings. Whereas distinguishing BD-I and BD-II main subtypes has a significant relevance for treatment strategy and for outcome, there are currently no clinical determinants of the BD subtype which could be used as early diagnostic predictors.

* While neurobiological specificity of each BD subtype is still controversial, available evidence suggest different dopaminergic abnormalities in each subtype. Dopaminergic function is involved in decision making and reward processing which may represent useful BD subtype markers.
* This study aims at assessing decision making during appetitive and punitive reinforcement learning in patients with BD I and BD II subtypes compared to healthy controls

ELIGIBILITY:
Inclusion Criteria:

* bipolar disorder (BD) type I or II, according to DSM (Diagnostic and Statistical Manual)-5 criteria
* Montgomery and Asberg Depression Rating Scale (MADRS) score < 15
* Young Mania Rating Scale (YMRS) score < 12

Exclusion Criteria:

* other main diagnosis than bipolar disorder
* other medical condition leading to cognitive deterioration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with bipolar disorder, type I and II, in a inter critical phase (euthymic period defined by the mood scales scores mentioned in the inclusion criteria)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-02-23 (Estimated); Study Completion 2022-02-23 (Estimated)

PRIMARY OUTCOMES:
Response performance in reward and loss trials | one day visit
  percentage of correct responses in the probabilistic learning task

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No